CLINICAL TRIAL: NCT07218471
Title: Prospective Changes in Patient-reported and Objective Functioning Following Reduction of Cannabis Use
Brief Title: Cannabis Reduction and Functional Outcomes
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rachel Tomko, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00145652; NIDA R01 DA062443 (Other Grant/Funding Number: National Institute on Drug Abuse (NIH/NIDA))
Record Dates: First submitted 2025-10-13; First posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Cannabis Use Disorder
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: CBT4CBT (Computerized Cognitive Behavioral Therapy) — Participants will receive one therapist-led motivational interviewing/goal setting session followed by 7 sessions of computerized CBT4CBT.
Behavioral: Motivational Interviewing — Participants will receive one therapist-led motivational interviewing/goal setting session followed by 7 sessions of computerized CBT4CBT.
Behavioral: Contingency Management — Patients will receive contingent reinforcers (financial incentives for reduction in urinary cannabinoids).

SUMMARY:
This study evaluates the effects of cannabis use reduction among adults diagnosed with cannabis use disorder (CUD). Participants will undergo an 8-week intervention combining motivational interviewing, computerized cognitive behavioral therapy (CBT4CBT), and financial incentives for reduction in urinary cannabinoids. The study aims to assess improvements in cannabis-related problems, sleep, cognitive performance, CUD severity, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Urinary cannabinoid level ≥ 50 ng/mL
* DSM-5 diagnosis of CUD (mild, moderate, or severe)
* Willingness to attempt cannabis reduction
* Completion of Intake Visit

Exclusion Criteria:

* Serious medical/psychiatric conditions
* Pregnancy or breastfeeding
* Use of cannabis in past 30 days was for medical purposes only
* Discontinuation or reduction of cannabis use may exacerbate a pre-existing condition
* TICS score ≤ 19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-09-15 (Estimated); Study Completion 2030-01-30 (Estimated)

PRIMARY OUTCOMES:
Cannabis-Related Problems | Week 8 (end-of-treatment)
  Rutgers Marijuana Problem Index (RMPI)- higher scores associated with worse outcomes.

SECONDARY OUTCOMES:
Total minutes of sleep per night | Week 8 (end-of-treatment)
  Measured via Fitbit Charge.
Minutes of light sleep per night | Week 8 (end-of-treatment)
  Measured via Fitbit Charge.
Minutes of rapid eye movement (REM) sleep per night | Week 8 (end-of-treatment)
  Measured via Fitbit Charge.
Minutes of deep sleep per night | Week 8 (end-of-treatment)
  Measured via Fitbit Charge.
Sleep efficiency rating | Week 8 (end-of-treatment)
  "Sleep score" as provided by Fitbit Charge. Range is 1-100 with higher scores indicating better sleep quality/efficiency.
Rey Auditory Verbal Learning Test (Verbal Memory) Age-Adjusted Standard Score | Week 8 (end-of-treatment)
  NIH Toolbox assessment; Higher scores indicate better cognitive functioning in this domain.
Face/Name Associative Memory Test (Visual Memory) Age-Adjusted Standard Score | Week 8 (end-of-treatment)
  NIH Toolbox assessment; Higher scores indicate better cognitive functioning in this domain.
Oral Symbol Digit Test Age-Adjusted Standard Score | Week 8 (end-of-treatment)
  NIH Toolbox assessment; Higher scores indicate better cognitive functioning in this domain.
Pattern Comparison Processing Speed Test (Processing Speed) Age-Adjusted Standard Score | Week 8 (end-of-treatment)
  NIH Toolbox assessment; Higher scores indicate better cognitive functioning in this domain.

OTHER OUTCOMES:
DSM-5 CUD Criteria and Severity | Week 8 (end-of-treatment)
  Clinician-administered semi-structured interview for assessing past month DSM-5 CUD symptoms
Quality of Life Enjoyment and Satisfaction-Q-SF | Week 8 (end-of-treatment)
  Self-report measure- range is 0-100% and higher percentages are associated with better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Tomko, PhD., Principal Investigator — Medical University of South Carolina; Erin McClure, PhD., Principal Investigator — Medical University of South Carolina